CLINICAL TRIAL: NCT00201422
Title: Eradication of Helicobacter Pylori in the Management of Stage IE & IIE-1 Primary Low-grade B Cell Lymphoma of Mucosa-associated Lymphoid Tissue Type of The Stomach
Brief Title: Eradication of Helicobacter Pylori in the Management of Stage IE & IIE-1 Primary Low-grade B Cell Lymphoma of MALToma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1296
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: MALT Lymphoma
Keywords: MALT lymphoma; diffuse large B-cell lymphoma,; stomach; Helicobacter pylori; antibiotic therapy
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse | interventions — Omeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omeprazole, Amoxicillin, Clarithromycin (Experimental): Anti-H. pylori Therapy (Triple therapy)
  Interventions: Other: Omeprazole, Amoxicillin, Clarithromycin

INTERVENTIONS:
Other: Omeprazole, Amoxicillin, Clarithromycin — Omeprazole20 mg,Clarithromycin500 mg b.i.d.,Day 1-14 plus Amoxicillin 500 mg q.i.d.,Day 1-14 plus

SUMMARY:
To evaluate the therapeutic effectiveness of H. pylori eradication in stage IE & IIE-1 primary low-grade B cell lymphoma of MALT of the stomach

DETAILED DESCRIPTION:
To investigate the prevalence of H. pylori infection in patients with early stage of primary low-grade B cell lymphoma of MALT of the stomach in Taiwan.

-To evaluate the therapeutic effectiveness of H. pylori eradication in stage IE & IIE-1 primary low-grade B cell lymphoma of MALT of the stomach.

To evaluate the efficacy of Helicobacter pylori eradication therapy with respect to objective regression rate and time to disease progression of primary low-grade gastric MALToma.

To estimate any differences in therapeutic efficacy related to different stage of disease,eg. stage IE v.s. stage IIE-1.

To identify the causes of treatment failure, such as the stage of tumor, the presence of large cell component, and/or persistent, reactivation or reinfection of H. pylori etc.

ELIGIBILITY:
Inclusion Criteria:

* The patients must have histologically confirmed primary low-grade B-cell lymphoma of MALT of the stomach which including the following types : diffuse small lymphocytic, diffuse small cleaved, and some diffuse mixed small and large cell types by Working Formulation (Harris NL et al. 1994)(20).
* The diagnosis of primary gastric lymphoma must fulfill the criteria of Dawson :

  1. No enlargement of peripheral or mediastinal lymph node;
  2. Peripheral blood smear revealing no leukemic or lymphomatous abnormalities;
  3. Predominant of alimentary tract lesions with any adenopathy corresponding to accepted lymphatic drainage route; and
  4. No involvement of liver or spleen except by extension of contiguous disease .
* The monoclonality of B-cell must be confirmed by either immunohisto- chemistry (light-chain restriction) or molecular technique (IgH rearrangement).
* The patient must have no prior chemotherapy or radiotherapy for his/her gastric MALToma.
* Patients must have evaluable disease by endoscopy and the nodal status by computed tomography. Endoscopic ultrasonography (EUS)* is optional and for reference only.
* H. pylori infection will be evaluated by the following tests: histology, rapid urease test (CLO-test), and serology C13-urea breath test (UBT) and bacterial culture* are optional and for reference only.
* The following will be considered to have H. pylori infection : at least two of the following 3 tests show positive results, rapid urease test (CLO-test), histology and serology.
* For C13-urea breath test, rapid urease test and histology to examine H. pylori, the examination must be performed at least 4 weeks apart from the latest antibiotics or non-steroid anti-inflammatory drug ingestion.
* Patients must have either stage IE or IIE-1 disease, according to an adaptation of the Ann Abor staging system modified by Musshoff for primary extranodal lymphoma.
* Stage IE : lymphoma confined to the gastric wall without lymph node involvement.
* Stage IIE : localized involvement of one or more GI site(s) on one side of the diaphragm with lymph node infiltration, any depth of lymphoma infiltration into the gut wall.
* Stage IIE-1 : infiltration of adjacent lymph node.
* Patient must have signed the informed consent.

Exclusion Criteria:

* Patients who have extensive gastrointestinal tract involvement are not eligible.
* Patients who have had previous history of extranodal lymphoma are not eligible.
* Patients who have disease beyond stage IIE-2: infiltration of regional lymph node, e.g. paraaortic, renal hilar, retroperitoneal, mesenteric, or lymph node of gastrosplenic ligment and of hepatoduodenal ligment are not eligible.
* Patients who had a history of allergic reaction to Amoxicillin and Erythromycin /Clarithromycin are not eligible.
* Patients whose cardiopulmonary status not allow him/her to have repeat endoscopy are not eligible.
* Patients who had prior surgery, chemo- or radiotherapy for their primary gastric lymphoma are not eligible.
* Patients who had previous anti-H. pylori therapy are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 1996-06; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy of Helicobacter pylori eradication therapy with respect to objective regression rate and time to disease progression of primary low-grade gastric MALToma. | Four weeks after the completion of anti-H. pylori therapy by CT scan
  Four weeks after the completion of anti-H. pylori therapy, patients shall have repeat endoscopy and abdominal CT to evaluate the H.pylori status and the response of MALToma.

SECONDARY OUTCOMES:
objective regression rate and time to disease progression of primary low-grade gastric MALToma. | 3-6 months by EUS
  atients who achieve complete or persistent partial response will receive no further treatment and have regular follow-up as section till tumor progression (relapse).

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, MD,PhD, Principal Investigator — Taiwan cooperative oncology group
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen LT, Lin JT, Tai JJ, Chen GH, Yeh HZ, Yang SS, Wang HP, Kuo SH, Sheu BS, Jan CM, Wang WM, Wang TE, Wu CW, Chen CL, Su IJ, Whang-Peng J, Cheng AL. Long-term results of anti-Helicobacter pylori therapy in early-stage gastric high-grade transformed MALT lymphoma. J Natl Cancer Inst. 2005 Sep 21;97(18):1345-53. doi: 10.1093/jnci/dji277. PMID 16174856
- See also: ISSN: 1460-2105, — http://english.nhri.org.tw/inst_cancer/ca_TCOGresearch.php